CLINICAL TRIAL: NCT03875898
Title: Study of the Impact of Daily Bread Consumption Enriched With a Fibre Mix on Intestinal Microbiota and Metabolic Profile in Subjects at Metabolic Risk
Brief Title: Bread Daily Intake Enriched With Mix Fibers in Metabolic Subjects: Intestinal Microbiota and Metabolic Profile Impact
Acronym: Breath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bridor (Industry)
Responsible Party: Principal Investigator, DUSSOUS Isabelle, Bridor Quality Manager, Bridor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Bridor
Record Dates: First submitted 2018-07-13; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Healthy Obesity, Metabolically
MeSH Terms: conditions — Obesity, Metabolically Benign

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 150 g bread fortified (15 g mix fibre) (Experimental): Volunteers will have to consume daily 150 g of a bread instead of usual bread during eight weeks
  Interventions: Other: 150 g bread fortified (15 g mix fibre)
- 150 g unfortified bread (Placebo Comparator): Volunteers will have to consume daily 150 g of an unfortified usual bread during eight weeks
  Interventions: Other: 150 g unfortified bread

INTERVENTIONS:
Other: 150 g bread fortified (15 g mix fibre) — Daily consumption of 150g of a bread fortified in fibre mix (15g) during eight weeks.
  Arms: 150 g bread fortified (15 g mix fibre)
Other: 150 g unfortified bread — Daily consumption of 150g of an usual bread in fibre-unfortified bread during eight weeks
  Arms: 150 g unfortified bread

SUMMARY:
The level of fibre consumption in France is lower than the national and international recommendations (mean 18.8 g/d for men, 16.4 g/d for women (INCA 2007 Study) instead of 30g/d recommended). Fibre have beneficial effects on health and interact with the intestinal microbiota diversity: a diet fortified with different structure fibres increase of 25 % the dysbiotic intestinal microbiota in obese patient (Cotillard et al, Dietary intervention impact on gut microbial gene richness. Nature, August 2013). The study aim is to evaluate the impact of daily consumption of bread (150 g ) enriched with a mixture of fibres of different structure (15g) during two months on the intestinal microbiota composition in metabolic risk subjects (abdominal overweight or obese) and also, to assess the correlation between the microbiota change and their metabolic profile improvement.It is a mono centric study with a centre in LYON (Centre de Recherche en Nutrition Humaine Rhône-Alpes)

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 25 to 35 kg/m2
* Waist circumference greater than 80 cm for women and than 96 cm for men
* Low level of fibre intake (<20 g /d) and low level of fibre nature diversity
* Daily bread consumption

Exclusion Criteria:

* Bread products allergy or intolerance
* Digestive surgery history except appendicectomy
* Metabolic or gastrointestinal disease history
* Medication that could interfere with glucose and lipid metabolism or intestinal microbiota (for example, no antibiotics within the 3 months before the study)
* Smokers (5 cig/d or more)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Intestinal microbiota composition at eight weeks | baseline and eight weeks
  intestinal microbiota composition will be measured by metagenomic analysis before all interventions, and before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)

SECONDARY OUTCOMES:
Change from baseline fasting and post prandial plasma glucose at eight weeks | baseline and eight weeks
  Plasma glucose will be measured in the fasting state and in the post-meal period over 7 hours before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)
Change from baseline fasting and post prandial plasma Insulin at eight weeks | baseline and eight weeks
  Plasma insulin will be measured in the fasting state and in the post-meal period over 7 hours before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)
Change from baseline fasting and post prandial plasma triglycerides at eight weeks | baseline and eight weeks
  Plasma triglycerides will be measured in the fasting state and in the post-meal period over 7 hours before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)
Change from baseline fasting and post prandial plasma non-esterified fatty acids at eight weeks | baseline and eight weeks
  Plasma non-esterified fatty acids will be measured in the fasting state and in the post-meal period over 7 hours before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)
Change from baseline fasting plasma lipids (cholesterol total, cholesterol HDL and LDL) at eight weeks | baseline and eight weeks
  Fasting plasma lipids will be measured before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)
Change from baseline C-Reactive Protein at eight weeks | baseline and eight weeks
  CRPus will be measured before and after each eight weeks, consumption sequences (fiber-fortified bread vs unfortified)
Change from baseline MDA (Malon Di Aldehyde) at eight weeks | baseline and eight weeks
  MDA will be measured before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)
Change from baseline Acetylated ghrelin at eight weeks | baseline and eight weeks
  Acylated ghrelin will be measured in the fasting state and postprandial period (at 0 and 240 min) before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)
Change from baseline Satiety evaluation at eight weeks | baseline and eight weeks
  Satiety response will be measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS) (on a 90mm horizontal line; from no sensation of satiety (minimal) to strong sensation of satiety (maximum).
Change from baseline Body composition at eight weeks | baseline and eight weeks
  Body composition will be measured with bio-impedancemetry before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified)
Change from Baseline Resting Energy Expenditure at eight weeks | baseline and eight weeks
  Resting Energy Expenditure will be measured with indirect calorimetry before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified).
Change from Baseline substrate oxydation at eight weeks | baseline and eight weeks
  Substrate oxydation (in the postprandial period over 7 hours) will be measured with indirect calorimetry before and after each eight weeks consumption sequence (fibre-fortified bread vs unfortified).
Change from baseline fibre intake at eight weeks | baseline and eight weeks
  The volunteers will complete a dietary survey of three days and fibre questionnaire
Change from baseline Gastrointestinal tolerance symptoms at eight weeks. | baseline and eight weeks
  Subjective ratings of bloating, nausea, vomiting, abdominal cramping and flatulence will be measured using visual analogue scale (VAS) score (on a 90mm horizontal line; from no symptom (minimal) to serious symptom (maximum).
Change from baseline stool consistency at eight weeks | baseline and eight weeks
  Stool consistency by Bristol Stool Chart (type1-7)

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, MD, Phd, Principal Investigator — Centre de Recherche en Nutrition Rhône-Alpes
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhône-Alpes, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website of the clinical investigation center — http://www.crnh-rhone-alpes.fr